CLINICAL TRIAL: NCT07132593
Title: A Retrospective, Observational, and Descriptive Study of Pediatric Cardiac Fibroma
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: T2024-ZX007-1
Record Dates: First submitted 2025-08-08; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Tumor
Keywords: congenital heart disease; cardiac tumor; surgical technique
MeSH Terms: conditions — Heart Neoplasms; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical group: Patients underwent cardiac fibroma resection and following ventricular reconstruction with the Sandwich Procedure.
  Interventions: Procedure: ventricular reconstruction

INTERVENTIONS:
Procedure: ventricular reconstruction — The Sandwich Procedure was developed at our institution to improve the strength and stability of heart wall reconstruction after tumor removal. It involves suturing two layers of treated biological tissue-both inside and outside the heart wall-to restore normal shape and function, while minimizing the risk of complications like aneurysm or bleeding.

SUMMARY:
This study was a retrospective descriptive case series analyzing outcomes of a novel surgical approach This study aimed to evaluate a modified surgical technique-called the Sandwich Procedure-for reconstructing the heart after resection of cardiac fibromas in children. Cardiac fibroma is a rare benign tumor that can compress vital cardiac structures and cause serious symptoms such as arrhythmia, heart failure, or obstruction of blood flow. Surgical removal is often required, but large tumors may leave defects in the heart wall that are challenging to repair, especially in young children.

The Sandwich Procedure was developed at our institution to improve the strength and stability of heart wall reconstruction after tumor removal. It involves suturing two layers of treated biological tissue-both inside and outside the heart wall-to restore normal shape and function, while minimizing the risk of complications like aneurysm or bleeding. This retrospective, observational study includes pediatric patients who underwent this procedure between 2018 and 2023. We report on its surgical feasibility, short- and mid-term outcomes, and potential benefits in preserving cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* underwent cardiac tumor resection
* underwent ventricular reconstruction with the Sandwich Procedure

Exclusion Criteria:

* the final pathological diagnosis indicated other than cardiac fibroma
* the final pathological diagnosis indicated metastatic tumors
* incomplete clinical or follow-up data

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients underwent cardiac fibroma resection followed by ventricular reconstruction with the Sandwich Procedure at our institution
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
composite endpoint | up to 5 years
  all-cause mortality or cardiac reoperation

SECONDARY OUTCOMES:
ventricular failure | up to 5 years
  left ventricular ejection fraction (LVEF) < 55% or right ventricular fractional area change (RVFAC) < 45% by echocardiography
ventricular aneurysm | up to 5 years
  newly formed segmental dyskinesia with localized dilation
malignant arrhythmia | up to 5 years
  sustained ventricular tachycardia, ventricular fibrillation, or frequent polymorphic premature ventricular contractions requiring medical intervention
Heart block | up to 5 years
  any new onset of high-degree atrioventricular block (Mobitz II or complete AVB), as well as complete left bundle branch block (CLBBB) by ECG
severe perioperative complications | before discharge
  including low cardiac output syndrome [cardiac index < 2.0 L/(min·m2)], delayed sternal closure, prolonged invasive mechanical ventilation (≥ 7 days) and need for extra-corporeal membrane oxygenation (ECMO)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Cardiac Surgery Center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data underlying this article cannot be shared publicly for the privacy of individuals that participated in the study.